CLINICAL TRIAL: NCT01077726
Title: A Single Arm, Open-label Trial Assessing the Effect of Capecitabine (Xeloda® ) on Progression-free Survival Rate at Four Months in Breast Cancer Patients With CNS Progression After Whole Brain Radiotherapy
Brief Title: A Study of Xeloda (Capecitabine) in Breast Cancer Patients With Central Nervous System (CNS) Progression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22203; 2008-007350-35
Record Dates: First submitted 2010-01-15; First posted 2010-03-01 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: capecitabine [Xeloda]

INTERVENTIONS:
Drug: capecitabine [Xeloda] — 1000mg/m2 po bid on days 1-14 of each 3 week cycle

SUMMARY:
This single arm study will assess the efficacy of Xeloda in the treatment of brain metastases in breast cancer patients with central nervous system (CNS) progression after whole brain radiotherapy. Patients will receive xeloda 1000mg/m2 po bid on days 1-14 of each 3 week cycle. The anticipated time on study treatment is until disease progression, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* female patients, >=18 years of age;
* breast cancer;
* CNS progression after radio-surgery + whole brain radiotherapy, or whole brain radiotherapy alone;
* at least one measurable lesion;
* ECOG performance status 0-2.

Exclusion Criteria:

* prior systemic treatment of brain metastases;
* prior disease progression while on Xeloda treatment;
* previous history of cancer (other than curatively treated basal and squamous cell cancer of the skin or in situ cancer of the cervix) in previous 5 years;
* clinically significant cardiovascular disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 4 months

SECONDARY OUTCOMES:
Objective Central Nervous System (CNS) response | From first administration of study treatment until documented CNS recurrence or progression
Duration of CNS response | From time of first documented cranial complete response (CR) or partial response (PR) (whichever is recorded first) until the first date CNS recurrence or progression is documented
Cranial PFS | From the first administration of study treatment to the time of documented cranial recurrence or progression\n
Progression-free survival\n | From the first administration of study treatment to the time of documented recurrence or progression\n
Clinical benefit \n | From first administration of study treatment to study end (12 Months)
Extra-cranial disease response rate\n | From first administration of study treatment to the time of documented extra-cranial recurrence or progression
Overall Survival (OS)\n | From first administration of study treatment to the time of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- France (11):
  - Angers
  - Arras
  - Béziers
  - Bobigny
  - Caen
  - Lille
  - Lyon
  - Narbonne
  - Nice
  - Paris
  - Salouël